CLINICAL TRIAL: NCT03505580
Title: Etude rétrospective et Prospective, Multicentrique, Non contrôlée, Non randomisée, Ouverte évaluant la Performance et la sécurité de l'Implant AMIStem
Brief Title: AMIStem-H Radiological Assessment
Status: Terminated | Type: Observational
Why Stopped: impossibility to carry on the study
Sponsor: Medacta International SA (Industry)
Responsible Party: Sponsor
Other Study IDs: P01.001.07
Record Dates: First submitted 2018-04-16; First posted 2018-04-23 (Actual); Last update posted 2025-09-29 (Actual); Status verified 2025-09

CONDITIONS: Hip Replacement Arthroplasty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | US Export: No

SUMMARY:
The purpose of this study is to evaluate radiological performance of the cementless femoral stem AMIStem H at 1 and 5-year follow-up.

All the patients operated at the investigational sites between April 2009 and April 2012 will be reviewed at 1, 5 and 10 year according to standard practice

ELIGIBILITY:
Inclusion Criteria:

* patients who underwent total hip arthroplasty at the investigational sites between April 2009 and April 2012
* patients bearing an AMIStem-H cementless femoral stem

Exclusion Criteria:

* patients who refuse to give consent for the treatment of data

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: All the patients who undewent total hip arthroplasty with AMIStem-H cementless femoral stem at the investigational sites between April 2009 and April 2012
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2013-10; Primary Completion 2022-12-31 (Actual); Study Completion 2025-08 (Actual)

PRIMARY OUTCOMES:
Presence of radiolucencies | 5 years

SECONDARY OUTCOMES:
correlation between the presence of radiolucencies and patient/implant characteristics | 5 years, 10 years
evaluation of radiolucent lines progression | 1 years, 10 years
evaluation of radiolucent lines progression | 5 years, 10 years
Record of adverse events | 1, 5 years and 10 years

CONTACTS AND LOCATIONS:
Locations (2):
- France (2):
  - Clinique Paris V, Paris, France
  - Clinique du Cèdre, Bois-Guillaume

IPD SHARING:
Plan to Share IPD: No